CLINICAL TRIAL: NCT00004047
Title: A Phase I Study of Intravenous DX-8951f in Patients With Advanced Myelodysplastic Syndromes, Refractory Acute Leukemia, Refractory or Transformed Chronic Lymphocytic Leukemia, and Chronic Myelogenous Leukemia in Blastic Phase
Brief Title: Chemotherapy in Treating Patients Who Have Hematologic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000067149; DAIICHI-8951A-PRT014; MDA-ID-99013; NCI-V99-1556
Record Dates: First submitted 1999-12-10; First posted 2004-07-19 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; blastic phase chronic myelogenous leukemia; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; chronic myelomonocytic leukemia; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Blast Crisis; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic | interventions — exatecan

INTERVENTIONS:
Drug: exatecan mesylate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of DX-8951f in treating patients who have hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of DX-8951f in patients with advanced myelodysplastic syndromes, refractory acute myeloid or lymphocytic leukemia, refractory or transformed chronic lymphocytic leukemia, or chronic myelogenous leukemia in blastic phase. II. Evaluate the quantitative and qualitative toxic effects of this regimen and determine the duration and reversibility of these effects in these patients. III. Make a preliminary determination of the antileukemic activity of this regimen in these patients. IV. Evaluate the pharmacokinetics of this regimen in these patients.

OUTLINE: This is a dose escalation study. Patients receive DX-8951f IV over 30 minutes daily for 5 days. Treatment continues every 3 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of DX-8951f until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose limiting toxicity. Patients are followed every 3 months until death.

PROJECTED ACCRUAL: Approximately 20-25 evaluable patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: One of the following hematologic malignancies: Advanced myelodysplastic syndromes Refractory anemia with excess blasts Refractory anemia with excess blasts in transformation Chronic myelomonocytic leukemia Refractory acute myeloid leukemia (AML) First salvage with primary refractory AML or first complete response (CR) no greater than 12 months in duration or at least second salvage therapy Once maximum tolerated dose is determined, intermediate AML prognosis (first CR duration greater than 12 months but less than 24 months) eligible Refractory acute lymphocytic leukemia Refractory or transformed chronic lymphocytic leukemia Chronic myelogenous leukemia in blastic phase No CNS disease

PATIENT CHARACTERISTICS: Age: Not specified Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: No specified Hepatic: Bilirubin no greater than 2.0 mg/dL SGOT or SGPT no greater than 2.0 times upper limit of normal Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No active congestive heart failure No uncontrolled angina No myocardial infarction within the past 6 months Other: Not pregnant or nursing Fertile patients must use effective contraception Negative pregnancy test No concurrent grade 4 infection No psychiatric disorder or mental disability No other life threatening illness

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent biologic therapy Chemotherapy: At least 30 days since prior cytotoxic therapy and recovered No concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: No concurrent radiotherapy to greater than 25% of skeleton Surgery: No concurrent surgery Other: At least 3 weeks since prior investigational drugs (including analgesics or antiemetics) Recovered from toxic effects of any prior therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-06; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L. DeJager, MD, FACP, Study Chair — Daiichi Sankyo
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Giles FJ, Cortes JE, Thomas DA, Garcia-Manero G, Faderl S, Jeha S, De Jager RL, Kantarjian HM. Phase I and pharmacokinetic study of DX-8951f (exatecan mesylate), a hexacyclic camptothecin, on a daily-times-five schedule in patients with advanced leukemia. Clin Cancer Res. 2002 Jul;8(7):2134-41. PMID 12114413